CLINICAL TRIAL: NCT02457611
Title: Open-Label Study to Evaluate the Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed-Dose Combination (FDC) for 6 Weeks in Subjects With Acute Genotype 1 or 4 Hepatitis C Virus (HCV) and Chronic Human Immunodeficiency Virus (HIV)-1 Co-Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed-Dose Combination (FDC) for 6 Weeks in Adults With Acute Genotype 1 or 4 Hepatitis C Virus (HCV) and Chronic Human Immunodeficiency Virus (HIV)-1 Co-Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1612; 2014-004812-12 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis C Infection With HIV Co-Infection
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDV/SOF (Experimental): LDV/SOF FDC for 6 weeks
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to determine the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in adults with acute genotype 1 or 4 hepatitis C virus (HCV) and chronic human immunodeficiency virus (HIV)-1 co-infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Acute, untreated, hepatitis C infection, genotype 1 or 4, with an estimated duration less than 24 weeks
* Confirmed HIV-1 infection
* CD4 T cell count >200/μL for individuals receiving antiretroviral therapy (ART), CD4 T cell count > 500/μL at screening for individuals without ART
* Use of two effective contraception methods if female of childbearing potential or sexually active male with female partner

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non HCV etiology
* Coinfection with hepatitis B virus (HBV)
* Treatment with any investigational drug or device within 60 days of the screening visit.
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- Germany (3):
  - Berlin
  - Bonn
  - Frankfurt am Main
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Rockstroh JK, Bhagani S, Hyland RH, Yun C, Dvory-Sobol H, Zheng W, Brainard DM, Ingiliz P, Lutz T, Boesecke C, Nelson M. Ledipasvir-sofosbuvir for 6 weeks to treat acute hepatitis C virus genotype 1 or 4 infection in patients with HIV coinfection: an open-label, single-arm trial. Lancet Gastroenterol Hepatol. 2017 May;2(5):347-353. doi: 10.1016/S2468-1253(17)30003-1. Epub 2017 Mar 1. PMID 28397698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany and the United Kingdom. The first participant was screened on 11 June 2015. The last study visit occurred on 8 January 2016.
Pre-assignment Details: 34 participants were screened.
Groups:
- LDV/SOF: Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet administered once daily for 6 weeks
Period: Overall Study
Arm/Group | LDV/SOF
Started | 26
Completed | 23
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- LDV/SOF: LDV/SOF 90/400 mg FDC tablet administered once daily for 6 weeks
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 24
  Asian | 1
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Not Disclosed | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 11
  Germany | 15
IL28b Status [Count of Participants; unit: Participants]
  CC | 12
  CT | 11
  TT | 3
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 19
  Genotype 4 | 7
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.4 (1.60)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 14
  >= 800,000 IU/mL | 12
CD4 Counts [Mean (Standard Deviation); unit: cells/uL] | 675 (251.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Completion of Treatment (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 1 or 4 HCV infection who were enrolled into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percentage of participants | 76.9 [56.4 to 91.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 6 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Discontinuation of Study Treatment (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after the last dose of study drug.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percentage of participants | 84.6 [65.1 to 95.6]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Weeks 2, 4, and 6
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percentage of participants
  Week 2 | 73.1 [52.2 to 88.4]
  Week 4 | 88.5 [69.8 to 97.6]
  Week 6 | 96.2 [80.4 to 99.9]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 2, 4, and 6
Time Frame: Baseline; Weeks 2, 4, and 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
log10 IU/mL
  Change at Week 2 | -4.01 (1.497)
  Change at Week 4: number analyzed (Participants) | 25
  Change at Week 4 | -4.16 (1.583)
  Change at Week 6: number analyzed (Participants) | 25
  Change at Week 6 | -4.17 (1.583)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure
    * confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment (ie, breakthrough),
    * confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment (ie, rebound),
    * HCV RNA persistently ≥ LLOQ through end of treatment (ie, nonresponse)
  * Relapse
    * HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percentage of participants | 15.4

7. Secondary Outcome: Change in HIV RNA From Day 1 to End of Treatment as Assessed by Proportion of Participants Who Had Confirmed HIV Virologic Rebound During the Study.
Description: Participants with HIV virologic rebound was defined as participants with at least two HIV RNA ≥ 400 copies/mL at 2 consecutive post-baseline visits which are at least 2 weeks apart based on actual dates.
Time Frame: Day 1; Week 6
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
Participants | 0

8. Secondary Outcome: Percentage of Participants That Maintain HIV-1 RNA < 50 Copies/mL While on HCV Treatment and at Posttreatment Week 4
Time Frame: Weeks 2, 4, 6, and Posttreatment Week 4
Population: Participants in the Safety Analysis Set who had HIV-1 RNA < 50 copies/mL at Baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 21
percentage of participants
  Week 2 | 100.0 [83.9 to 100.0]
  Week 4 | 100.0 [83.9 to 100.0]
  Week 6 | 95.2 [76.2 to 99.9]
  Posttreatment Week 4 | 100.0 [83.9 to 100.0]

9. Secondary Outcome: Percent Change From Baseline in CD4 T-cell Count at the End of Treatment and at Posttreatment Week 4
Time Frame: Baseline; Week 6; Posttreatment Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LDV/SOF
Number analyzed (Participants) | 26
percent change
  Change at Week 6: number analyzed (Participants) | 24
  Change at Week 6 | -0.3 (4.91)
  Change at Posttreatment Week 4: number analyzed (Participants) | 23
  Change at Posttreatment Week 4 | 0.4 (4.08)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=26)
Pyrexia (General disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=26)
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 2
Syphilis (Infections and infestations) | 2
Headache (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 3

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years